CLINICAL TRIAL: NCT02395666
Title: A Phase II Preventative Trial of DFMO (Eflornithine HCl) as a Single Agent in Patients With High Risk Neuroblastoma in Remission
Brief Title: Preventative Trial of Difluoromethylornithine (DFMO) in High Risk Patients With Neuroblastoma That is in Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Giselle Sholler (Other)
Collaborators: Beat NB Cancer Foundation (Other); Because of Ezra (Other); K C Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor-Investigator, Giselle Sholler, Beat Childhood Cancer Chair, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NMTRC003B; NCT01586260 (obsolete NCT alias)
Record Dates: First submitted 2015-03-05; First posted 2015-03-23 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma in remission; Relapsed Neuroblastoma; Refractory Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Eflornithine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DFMO twice daily (Experimental): Subjects will receive twenty-seven (27) cycles of oral DFMO at a dose of 500 to 1000 mg/m2 BID on each day of a 28 day cycle.
  Interventions: Drug: DFMO

INTERVENTIONS:
Drug: DFMO — Subjects will receive twenty-seven (27) cycles of oral DFMO at a dose of 500 to 1000 mg/m2 BID on each day of a 28 day cycle.
  Other Names: eflornithine HCl; Difluoromethylornithine

SUMMARY:
The purpose of this research study is to evaluate a new investigational drug to prevent reoccurrence of neuroblastoma that is in remission. This study drug is called DFMO. The objectives of this study will be to monitor for safety and look at efficacy of DFMO.

The safety of the proposed dosing regimen in this trial will be tested by an on-going risk/benefit assessment during the study. A patient benefiting from treatment, not progressing on therapy, and in the absence of any safety issues associated with DFMO may continue on treatment up to 27 cycles with the expectation that there will be an overall clinical benefit.

The procedures involved in this study include Medical history, Physical exam, Vital signs (blood pressure, pulse, temperature), Blood tests, Urine tests, MRI or CT scan of the tumor(s), meta-iodobenzylguanidine (MIBG) scans, and Bone marrow aspirations. All of these tests and procedures are considered standard of care for this population. Drug administration is also part of this protocol, including an investigational new drug called DFMO.

The proposed dosing regimen is an oral dose of DFMO tablets two times a day for each day while on study. There will be 27 cycles. Each cycle will be 28 days in length.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0-21 years at the time of diagnosis.
* Diagnosis: histologic verification at either the time of original diagnosis or a previous relapse of high risk neuroblastoma.
* Disease Status: Neuroblastoma that is in remission
* First dose of study medication must be greater than 30 days from completion of cytotoxic and antibody therapy and less than 120 days from previous therapy
* A negative serum or urine pregnancy test is required for female subjects of child bearing potential (onset of menses or ≥13 years of age).
* Both male and female post-pubertal study subjects need to agree to use one of the more effective birth control methods during treatment and for six months after treatment is stopped. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonorgestrel implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
* Absolute Neutrophil Count (ANC) > 500/μl and platelet count >50,000/μl
* Organ Function Requirements: Subjects must have adequate liver function as defined by:

  * Aspartate Aminotransferase (AST) and Alanine transaminase (ALT) <10x upper limit of normal
  * Serum bilirubin must be ≤ 2.0 mg/dl
  * Serum creatinine based on age/gender
* Informed Consent: All subjects and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

* Lansky score < 60%
* Body Surface Area (BSA) (m2) of <0.25
* Investigational Drugs: Subjects who are currently receiving another investigational drug are excluded from participation.
* Anti-cancer Agents: Subjects who are currently receiving other anticancer agents are not eligible. Subjects must have fully recovered from the effects of prior chemotherapy (hematological and bone marrow suppression effects).
* Infection: Subjects who have an uncontrolled infection are not eligible until the infection is judged to be well controlled in the opinion of the investigator.
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study, or in whom compliance is likely to be suboptimal, should be excluded.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2015-03-05 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2023-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Saulnier-Sholler, MD, Study Chair — Beat Childhood Cancer
Locations (22):
- United States (22):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Rady Children's Hospital, San Diego, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - All Children's Hospital Johns Hopkins Medicine, St. Petersburg, Florida
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tufts Medical Center, Boston, Massachusetts
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospital and Clinics on Minnesota, Minneapolis, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center and Children's Hospital, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Monroe Carrell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Dell Children's Blood and Cancer Center, Austin, Texas
  - Children's Medical Center, Dallas, Texas
  - Texas Children's Cancer and Hematology Centers, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah

REFERENCES:
- [Derived] Duke ES, Bradford D, Sinha AK, Mishra-Kalyani PS, Lerro CC, Rivera D, Wearne E, Miller CP, Leighton J, Sabit H, Zhao H, Lane A, Scepura B, Pazdur R, Singh H, Kluetz PG, Donoghue M, Drezner N. US Food and Drug Administration Approval Summary: Eflornithine for High-Risk Neuroblastoma After Prior Multiagent, Multimodality Therapy. J Clin Oncol. 2024 Sep 1;42(25):3047-3057. doi: 10.1200/JCO.24.00546. Epub 2024 Jun 25. PMID 38917371
- [Derived] Oesterheld J, Ferguson W, Kraveka JM, Bergendahl G, Clinch T, Lorenzi E, Berry D, Wada RK, Isakoff MS, Eslin DE, Brown VI, Roberts W, Zage P, Harrod VL, Mitchell DS, Hanson D, Saulnier Sholler GL. Eflornithine as Postimmunotherapy Maintenance in High-Risk Neuroblastoma: Externally Controlled, Propensity Score-Matched Survival Outcome Comparisons. J Clin Oncol. 2024 Jan 1;42(1):90-102. doi: 10.1200/JCO.22.02875. Epub 2023 Oct 26. PMID 37883734
- [Derived] Urban-Wojciuk Z, Graham A, Barker K, Kwok C, Sbirkov Y, Howell L, Campbell J, Woster PM, Poon E, Petrie K, Chesler L. The biguanide polyamine analog verlindamycin promotes differentiation in neuroblastoma via induction of antizyme. Cancer Gene Ther. 2022 Jul;29(7):940-950. doi: 10.1038/s41417-021-00386-6. Epub 2021 Sep 14. PMID 34522028
- [Derived] Batth IS, Dao L, Satelli A, Mitra A, Yi S, Noh H, Li H, Brownlee Z, Zhou S, Bond J, Wang J, Gill J, Sholler GS, Li S. Cell surface vimentin-positive circulating tumor cell-based relapse prediction in a long-term longitudinal study of postremission neuroblastoma patients. Int J Cancer. 2020 Dec 15;147(12):3550-3559. doi: 10.1002/ijc.33140. Epub 2020 Jun 23. PMID 32506485
- [Derived] Lewis EC, Kraveka JM, Ferguson W, Eslin D, Brown VI, Bergendahl G, Roberts W, Wada RK, Oesterheld J, Mitchell D, Foley J, Zage P, Rawwas J, Rich M, Lorenzi E, Broglio K, Berry D, Saulnier Sholler GL. A subset analysis of a phase II trial evaluating the use of DFMO as maintenance therapy for high-risk neuroblastoma. Int J Cancer. 2020 Dec 1;147(11):3152-3159. doi: 10.1002/ijc.33044. Epub 2020 May 24. PMID 32391579
- See also: Beat Childhood Cancer Consortium website — http://www.beatcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Stratum 1: Subjects that are in remission at the end of upfront therapy defined as chemotherapy (5-7 cycles), surgery as indicated, consolidation therapy as indicated, radiation therapy as indicated, anti-GD2 antibody therapy with retinoic acid up to 6 cycles.
  Subjects will receive twenty-seven (27) cycles of oral DFMO at a dose of 500 to 1000 mg/m2 BID on each day of a 28 day cycle.
- Stratum 2: Subjects that are in remission after any previous relapse or refractory therapy.
  Subjects will receive twenty-seven (27) cycles of oral DFMO at a dose of 500 to 1000 mg/m2 BID on each day of a 28 day cycle.
Period: Overall Study
Arm/Group | Stratum 1 | Stratum 2
Started | 101 | 39
Completed | 95 | 38
Not Completed | 6 | 1
Not completed — Physician Decision | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 | Stratum 2 | Total
Number analyzed (Participants) | 101 | 39 | 140
Age, Continuous [Mean (Full Range); unit: years] | 4.4 [1 to 17] | 6.8 [1 to 14] | 5.1 [1 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 11 | 55
  Male | 57 | 28 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 82 | 32 | 114
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Event Free Survival (EFS) During Study.
Description: To evaluate the preventative activity of DFMO as a single agent in patients that are in remission based on: Event free survival (EFS)
Time Frame: 2 Years
Population: One subject removed from Stratum 1 due to not fitting study criteria upon review
Measure: Mean (95% Confidence Interval); unit: percentage of subjects without an event
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 100 | 39
percentage of subjects without an event | 84 [80 to 88] | 51 [43 to 59]

2. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: To evaluate the preventative activity of DFMO as a single agent in patients with neuroblastoma who are in remission based on: Overall Survival (OS)
Time Frame: 2 Years
Measure: Mean (95% Confidence Interval); unit: percentage of subjects without an event
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 100 | 39
percentage of subjects without an event | 97 [95 to 99] | 84 [78 to 90]

3. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: To continue to determine the safety and tolerability of DFMO as a single agent and in pediatric and young adult patients with high risk neuroblastoma that is in remission.
Time Frame: 2 years
Population: Stratum 1 and 2 were analyzed together as one safety group as per statistical analysis plan.
Measure: Count of Participants; unit: Participants
Arm/Group | DFMO Twice Daily
Number analyzed (Participants) | 140
Participants | 57

4. Secondary Outcome: Test the Association of Survival With ODC1 Genotype
Description: Tests (p-value) of the association of survival with ODC1 single nucleotide polymorphism rs2302616 genotype.
  Blood: microRNA analysis as predictor of DFMO effect, ornithine decarboxylase (ODC) single nucleotide polymorphism (SNP) analysis in DNA isolated from nucleated cells
Time Frame: 2 years
Population: Stratum 1 and 2 were analyzed together as one group as per statistical analysis plan.
Measure: Number; unit: p-value
Groups:
- GG, GT, TT; GG or GT, TT; GG, GT or TT: Tests of the association of survival with ODC1 single nucleotide polymorphism rs2302616 genotype.
Arm/Group | GG, GT, TT | GG or GT, TT | GG, GT or TT
Number analyzed (Participants) | 140 | 140 | 140
p-value | 0.96 | 0.58 | 0.67

5. Secondary Outcome: Peak Plasma Concentration (Cmax)
Description: Pharmacokinetic assay Cmax/D
  Samples drawn at 5 timepoints: (0 (pre dose), 30min, 1 hour, 3 hours, and 6 hours post-dose) on two different days.
Time Frame: Samples drawn at 5 timepoints: (0 (pre dose), 30min, 1 hour, 3 hours, and 6 hours post-dose) on two different days
Population: 12 subjects from both Stratum 1 and 2 were analyzed together as one group as per statistical analysis plan.
Measure: Mean (90% Confidence Interval); unit: ng/mL
Groups:
- Study Subjects Consented to PK Collection: Includes study subjects from either stratum that signed an optional consent to have PK's collected
Arm/Group | Study Subjects Consented to PK Collection
Number analyzed (Participants) | 12
ng/mL | 11958 [5123 to 18793]

6. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC)
Description: Pharmacokinetic assay AUC(0-6 hr)/D
  Samples drawn at 5 timepoints: (0 (pre dose), 30min, 1 hour, 3 hours, and 6 hours post-dose) on two different days
Time Frame: 0 (pre dose), 30min, 1 hour, 3 hours, and 6 hours post-dose on two different days
Population: 12 subjects from both Stratum 1 and 2 were analyzed together as one group as per statistical analysis plan.
Measure: Mean (90% Confidence Interval); unit: hr*ng/mL
Arm/Group | Study Subjects Consented to PK Collection
Number analyzed (Participants) | 12
hr*ng/mL | 47024 [23868 to 70180]

7. Secondary Outcome: Time to Reach Peak Plasma Concentration (Tmax)
Description: Pharmacokinetic assay- tmax, hr
  Samples drawn at 5 timepoints: (0 (pre dose), 30min, 1 hour, 3 hours, and 6 hours post-dose) on two different days
Time Frame: 0 (pre dose), 30min, 1 hour, 3 hours, and 6 hours post-dose on two different days
Population: 12 subjects from both Stratum 1 and 2 were analyzed together as one group as per statistical analysis plan.
Measure: Mean (90% Confidence Interval); unit: hours
Arm/Group | Study Subjects Consented to PK Collection
Number analyzed (Participants) | 12
hours | 3.3 [1.9 to 4.7]

ADVERSE EVENTS:
Time Frame: Through study completion plus 30 days, an average of 2 years.
Description: All subjects that received at least one dose of DFMO. Since both arms received the same exact treatment, they were combined into one reporting group.
Groups:
- All Study Subjects: All subjects that received at least one dose of DFMO. Since both arms received the same exact treatment, they were combined into one reporting group.
Arm/Group | All Study Subjects
All-Cause Mortality (participants affected / at risk) | 0/140
Serious Adverse Events (participants affected / at risk) | 23/140
Other Adverse Events (participants affected / at risk) | 41/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Subjects (N=140)
Infection (Infections and infestations) | 8 (8) — All Unrelated
Vomiting (Gastrointestinal disorders) | 3 (3) — All Unrelated
Pain (General disorders) | 1 (1) — Unrelated
Diarrhea (Gastrointestinal disorders) | 3 (3) — All Unrelated
Fever (General disorders) | 1 (1) — Unrelated
Hyponatremia (Investigations) | 1 (1) — Unrelated
Benign vascular lesion (Vascular disorders) | 1 (1) — Unrelated
Swelling of Eye (Eye disorders) | 1 (1) — Eye swelling result of brain mass that has been confirmed as metastatic recurrent neuroblastoma. Unrelated
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) — Possibly related
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) — Possibly related
Constipation (Gastrointestinal disorders) | 1 (1) — Unrelated
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Unrelated
Hypotension (Cardiac disorders) | 1 (1) — Unrelated
hearing loss (Ear and labyrinth disorders) | 1 (1) — Possibly related
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Femur Fracture- Unrelated
Influenza (Infections and infestations) | 1 (1) — Unrelated
Bacteremia (Infections and infestations) | 1 (1) — Unrelated
Obstruction (Gastrointestinal disorders) | 1 (1) — gastric obstruction secondary to adhesions from previous surgery. Resolved after surgical correction. Unrelated
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Subjects (N=140)
Neutrophil count decrease (Blood and lymphatic system disorders) | 11 (11)
Anemia (Blood and lymphatic system disorders) | 6 (6)
ALT elevation (Hepatobiliary disorders) | 14 (14)
AST elevation (Hepatobiliary disorders) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Hearing Loss (Ear and labyrinth disorders) | 9 (9)
Otitis Media (Infections and infestations) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-18): https://cdn.clinicaltrials.gov/large-docs/66/NCT02395666/Prot_SAP_001.pdf